CLINICAL TRIAL: NCT01768520
Title: For 12 Weeks, the Multi-center, Randomized, Double-blinded, Clinical Study to Evaluate the Efficacy and Safety of Entelon Tab. 150mg Compared With Celebrex Capsule in Patients With Osteoarthritis of Knee (Phase III)
Brief Title: Evaluation of the Efficacy and Safety of Entelon Tab. 150mg in Patients With Osteoarthritis of Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HL_ENTR_302
Record Dates: First submitted 2013-01-14; First posted 2013-01-15 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — whole grape extract; Celecoxib; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Entelon tab. 150mg (Experimental)
  Interventions: Drug: Enteron tab. 150mg(vitis vinifera extract 150mg) : twice daily for 12 weeks
- Celebrex cap. (Active Comparator)
  Interventions: Drug: Celebrex cap. (celecoxib 200mg) : once daily, for 12 weeks
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enteron tab. 150mg(vitis vinifera extract 150mg) : twice daily for 12 weeks — 1. morning : 1 tab. of active Entelon 150mg plus 1 cap. of placebo Celebrex
  2. evening : 1 tab. of active Entelon 150mg
  Arms: Entelon tab. 150mg
Drug: Celebrex cap. (celecoxib 200mg) : once daily, for 12 weeks — 1. morning : 1 tab. of placebo Entelon 150mg + 1 cap. of active Celebrex
  2. evening : 1 tab. of placebo Entelon 150mg
  Arms: Celebrex cap.
Drug: Placebo — 1. morning : 1 tab. of placebo Entelon 150mg + 1 cap. of placebo Celebrex
  2. evening : 1 tab. of placebo Entelon 150mg
  Arms: Placebo

SUMMARY:
This clinical trial is planned to prove Entelon tab. arm is not inferior to Celebrex cap. arm in terms of the efficacy and safety through the change of K-WOMAC's total score sum in patients with osteoarthritis of knee.

ELIGIBILITY:
Inclusion Criteria:

1. both gender,35 years ≤ age ≤ 75 years
2. patients with a diagnosis of OA(osteoarthritis) of the knee within 3 months prior to study participation, as determined by the American College of Rheumatology clinical and radiographic criteria as follows.

   1. knee arthralgia
   2. more than one case among

      * 50 years or over

        * morning stiffness less than 30 min

          * friction sound
   3. osteophyte in radiography
3. Kellgren and Lawrence Scale Grade II~III
4. total sum of K-WOMAC Scale more than 30
5. negative results in pregnancy test of urine in screening period
6. if women in childbearing age, medically reliable contraception or menopause
7. patients who give written consent of agreement to voluntarily participate in the clinical study
8. patients who can read and understand written instructions

Exclusion Criteria:

1. patients whose total sum of K-WOMAC in visit 2 is less than that in visit 1
2. fibromyalgic, anserine bursitis, infectious arthritis, rheumatoid arthritis, ankylosing spondylitis, gout or pseudogout
3. knee OA with secondary causes including major dysplastic or congenital malformation, ochronosis, acromegaly, Hemochromatosis, Wilson's disease or primary osteochondromatosis
4. anatomical malformation, disease of vertebra or other lower extremities or other disease of orthopedics which can disturb the evaluation of the target joint
5. wound, inflammation or avascular necrosis of the target joint or arthroscopy within 6 months prior to study participation
6. patients with administration of injectable hyaluronic acid to the target joint within 6 months prior to study participation
7. severe ischaemic heart diseases, peripheral artery disease and/or cerebrovascular disease, congestive heart failure, active bronchial asthma
8. medical history of malignant tumor
9. active peptic ulcer, gastrointestinal tract bleeding or inflammatory bowel disease
10. hypersensitivity with aspirin, celecoxib, corticosteroid, acetaminophen, sulfonamide derivatives or vitis vinifera or intolerance with fructose, glucose or galactose
11. continuously(1 week or more) oral or intraarticular administration of corticosteroids within 12 weeks prior to study participation
12. pregnant or lactating women
13. patients who have experience to participate in other clinical trial within 4 weeks prior to study participation
14. ALT, AST and Serum Creatinine ≥ 2×UNL
15. drug administration after diagnosing as alcoholic or psychical disease
16. patients whom the investigators judge as improper to participate in this clinical trial

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2012-07-02 (Actual); Primary Completion 2014-10-15 (Actual); Study Completion 2015-05-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Kyoung-gi Do, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Entelon Tab. 150mg | Celebrex Cap. | Placebo
Started | 152 | 147 | 39
Completed | 120 | 121 | 30
Not Completed | 32 | 26 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entelon Tab. 150mg | Celebrex Cap. | Placebo | Total
Number analyzed (Participants) | 152 | 147 | 39 | 338
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.41 (7.41) | 62.24 (7.12) | 64.13 (6.76) | 62.09 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 105 | 31 | 260
  Male | 28 | 42 | 8 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 152 | 147 | 39 | 338
Part of Osteoarthritis diagnosis [Number; unit: participants]
  Right knee | 72 | 70 | 17 | 159
  Left knee | 80 | 77 | 22 | 179

OUTCOME MEASURES:

1. Primary Outcome: the Change of Total Sum of K-WOMAC(Korean The Western Ontario and McMaster Universities Arthritis Index)
Description: Range of total K-WOMAC score: 0-96 K-WOMAC consists of evaluations of pain, stiffness, physical function. The total K-WOMAC score is the sum of all subscale scores. Higher scores mean a worse outcome.
  Range of Subscale K-WOMAC score: pain(0-20), stiffness(0-8), physical function(0~68) Higher scores mean a worse outcome.
  If there is missing data, LOCF(Last Observation Carried Forward) was applied and analyzed.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Entelon Tab. 150mg | Celebrex Cap. | Placebo
Number analyzed (Participants) | 120 | 121 | 30
score on a scale
  baseline | 51.64 (13.62) | 54.57 (14.06) | 49.94 (11.81)
  12 weeks | 30.68 (18.69) | 33.88 (20.44) | 33.80 (15.98)
  change(12 weeks-baseline) | -19.38 (19.79) | -19.26 (18.22) | -16.70 (20.10)

2. Secondary Outcome: the Change of Numeric Rating Scale
Description: Numeric Rating Scale is 10 point scale(0~10 score). 0 score: no pain, 10 score: worst possible pain
  If there is missing data, LOCF(Last Observation Carried Forward) was applied and analyzed.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Entelon Tab. 150mg | Celebrex Cap. | Placebo
Number analyzed (Participants) | 120 | 121 | 30
score on a scale
  baseline | 5.62 (1.40) | 5.54 (1.73) | 5.44 (1.67)
  12 weeks | 3.57 (2.07) | 4.09 (2.09) | 4.23 (2.22)
  change(12weeks-baseline) | -2.14 (1.81) | -1.54 (2.34) | -1.50 (1.86)

ADVERSE EVENTS:
Time Frame: 12Weeks
Arm/Group | Entelon Tab. 150mg | Celebrex Cap. | Placebo
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/147 | 0/39
Serious Adverse Events (participants affected / at risk) | 3/152 | 4/147 | 1/39
Other Adverse Events (participants affected / at risk) | 14/152 | 22/147 | 16/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entelon Tab. 150mg (N=152) | Celebrex Cap. (N=147) | Placebo (N=39)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nasolacrimal duct obstruction,Right (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Middle cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
three abscess cavities scattered in both hepatic lobes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Entelon Tab. 150mg (N=152) | Celebrex Cap. (N=147) | Placebo (N=39)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes